CLINICAL TRIAL: NCT04200365
Title: A Pilot Study of INCB039110 (Itacitinib) for the Treatment of Steroid Refractory Chronic Graft-Versus-Host Disease
Brief Title: A Study of Itacitinib for the Treatment of Chronic Graft Versus Host Disease (cGVHD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment and PI departure
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT29
Record Dates: First submitted 2019-12-10; First posted 2019-12-16 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-08

CONDITIONS: Chronic Graft-versus-host-disease
Keywords: Chronic Graft-versus-host-disease; Allogeneic hematopoietic stem cell transplant; Corticosteroids; Immunosuppressive therapies
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — itacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Itacitinib (Experimental)
  Interventions: Drug: Itacitinib

INTERVENTIONS:
Drug: Itacitinib — Itacitinib will be administered orally once daily for up to 24 months.
  Other Names: INCB039110 adipate

SUMMARY:
This study is being done in patients who have been receiving corticosteroids or other immunosuppressive therapies for the treatment of cGVHD for at least 6 months. The purpose of this study is to find out if itacitinib in combination with corticosteroids or other immunosuppressive therapies is safe and effective in people with cGVHD.

DETAILED DESCRIPTION:
Graft versus host disease remains a major hurdle to improve allogeneic hematopoietic stem cell transplantation outcome, with cGVHD being associated with decreased quality of life. Suppression of the immune system with corticosteroids forms the basis of first-line therapy for management of GVHD, but sustained responses are usually seen in less than 50 percent of patients and there is no standard second- or third-line treatment for steroid refractory cGVHD. Identification of novel therapeutic targets are needed to improve outcomes. Therapeutic potential has been shown by a JAK inhibitor in the treatment of steroid refractory GVHD. Itacitinib is a novel, selective inhibitor of the JAK family of protein tyrosine kinases and will be studied here in patients with steroid refractory cGVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed by the patient or legal guardian prior to any study-related screening procedures
2. Patients who have undergone allo-hematopoietic stem cell transplant(s) (HSCT) from any donor HLA type (related or unrelated donor with any degree of HLA matching) using any graft source (bone marrow, peripheral blood stem cells, or cord blood). Recipients of non-myeloablative, myeloablative, and reduced intensity conditions are eligible.
3. Active, clinically diagnosed, moderate or severe cGVHD per NIH Consensus Criteria:

   * Moderate cGVHD: at least 1 organ (except lung) with a score of 2, ≥3 organs involved with a score of 1 in each organ, or lung score of 1
   * Severe cGVHD: at least 1 organ with a score of 3, or lung score of 2 or 3
4. cGVHD must be refractory to steroids defined by at least one criteria:

   * Patient is refractory to glucocorticoid therapy at screening: ongoing treatment with prednisone equivalent ≥0.20 mg/kg/day x 4 weeks (wks) at screening and organ progression documented 4 wks after the initiation of this regimen
   * Patient is dependent on glucocorticoid therapy at screening: treatment with a prednisone equivalent mean dose ≥0.20 mg/kg/day received for 12 wks at screening
   * Patient is intolerant to glucocorticoids at screening: ongoing treatment with prednisone equivalent ≥0.20 mg/kg/day x 4 wks at screening and presence of at least one documented glucocorticoid toxicity
5. Evidence of myeloid and platelet engraftment (absolute neutrophil count ˃1,000/mm^3 and platelet count ˃25,000/mm^3). Use of growth factors or platelet transfusions is not allowed within 7 days before screening of laboratory assessment.
6. Patients must currently be receiving systemic or other immunosuppressive therapies for the treatment of cGVHD for a duration of ˃6 months prior to start of study treatment
7. Patients must be able to swallow and retain oral medication
8. Eastern Cooperative Oncology Group Performance Status score of 0, 1, or 2
9. Adequate hematologic function
10. Adequate renal function: creatinine clearance ≥30 mL/min measured or calculated by Cockcroft Gault equation
11. Patients willing to avoid pregnancy or father children based on 1 of the following:

    * Women of non-childbearing potential (i.e., surgically sterile by hysterectomy and/or bilateral oophorectomy OR ≥12 months of amenorrhea)
    * Women of childbearing potential who have a negative serum pregnancy test at screening and who agree to take appropriate precautions to avoid pregnancy from screening through safety follow-up.
    * Men who agree to take appropriate precautions to avoid fathering children from screening through safety follow-up. Male patients must also refrain from donating sperm during their participation in the study and for at least 3 months after completing the study.
12. Ability to understand the nature of this study and to comply with study and follow-up procedures

Exclusion Criteria:

1. Receiving concomitant JAK inhibitor for cGVHD; prior treatment with a JAK inhibitor for acute GVHD is permitted if treatment was stopped more than 60 days prior to study start. Patients are eligible if JAK inhibitors for treatment of cGVHD are stopped due to side effects and not due to refractoriness.
2. Treatment with any other investigational agent, device, or procedure, within 28 days (or 5 half-lives, whichever is longer) of enrollment. For previous study drugs where 5 half-lives is ≤28 days, a minimum of 10 days between termination of that study drug and administration of itacitinib is required.
3. Presence of current secondary malignancies with the exception of previously treated in situ carcinoma, cervical carcinoma Stage 1B or less, and noninvasive basal cell or squamous cell skin carcinoma.
4. Pregnant or nursing (lactating) women
5. Patients with relapsed primary malignancy, or who have been treated for relapse after the allo-HSCT was performed
6. History of progressive multifocal leukoencephalopathy
7. Evidence of the following infections:

   * Active uncontrolled bacterial, fungal, parasitic, or viral infection. Infections are considered controlled if appropriate therapy has been instituted and, at the time of screening, no signs of infection progression are present. Progression of infection is defined as hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
   * Known HIV infection
   * Active tuberculosis infection that developed after allo-HSCT
   * Active viral infection confirmed by polymerase chain reaction for the BK virus ( a polyoma virus), cytomegalovirus, Epstein-Barr virus, and human herpes virus 6
   * Active hepatitis B virus (HBV) or hepatitis C virus that requires treatment, or at risk for HBV reactivation (i.e., positive HBsAg)
8. Severe organ dysfunction unrelated to underlying GVHD including:

   * Cholestatic disorders or unresolved veno-occlusive disease of the liver (persistent bilirubin abnormalities not attributable to GVHD and ongoing organ dysfunction)
   * Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral itacitinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowl resection)
   * Clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial infarction within 6 months of enrollment, New York Heart Association Class III or IV congestive heart failure, circulatory collapse requiring vasopressor or inotropic support, or arrhythmia that requires therapy
   * Significant respiratory disease that requires mechanical ventilation support or a resting O2 saturation ˂90 percent by pulse oximetry or FEV1 ˂30 percent
9. Patients requiring platelet transfusions to maintain a platelet count ˃25,000/mm^3
10. Any corticosteroid therapy for indications other than cGVHD at doses ˃1 mg/kg/day methylprednisone or equivalent within 7 days of study start
11. Patients receiving treatment with medications that interfere with coagulation or platelet function including, but not limited to, aspirin dose exceeding 81 mg/day and related drugs such as heparin or warfarin sodium. Use of low molecular weight heparin is allowed.
12. Known allergies, hypersensitivity, or intolerance to itacitinib or any of its excipients
13. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - South Austin Medical Center, Austin, Texas
  - Texas Oncology - Sammons Cancer Center, Dallas, Texas
  - Texas Transplant Institute, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Itacitinib
Started | 15
Completed | 4
Not Completed | 11
Not completed — Adverse Event | 2
Not completed — Progressive Disease | 4
Not completed — Lack of Efficacy | 1
Not completed — Study Closure | 4

BASELINE CHARACTERISTICS:
Groups:
- Itacitinib: Itacitinib: Participants received itacitinib orally once daily for up to 24 months.
Arm/Group | Itacitinib
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 59.5 [27 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: cGVHD Overall Response Rate (ORR) at 6 Months on Treatment
Description: Defined as the rate of participants with a cGVHD response of complete response (CR) or partial response (PR) after 6 months of treatment with Itacitinib as defined by 2014 National Institutes of Health Consensus Development Project on Clinical Trials in cGVHD. CR is defined as resolution of all manifestations of cGVHD in each organ or site. PR is defined as the improvement in at least one organ or site without progression in any other organ or site.
Time Frame: Response assessed Day 1 of every cycle up until the end of treatment, up to 24 months. This outcome measure is the ORR for all patients once they have been on treatment for 6 months.
Population: Participants must have had one dose of study drug and must have had 1 post-baseline disease evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Itacitinib
Number analyzed (Participants) | 15
percentage of participants | 93

2. Secondary Outcome: Number of Participants That Can Withdraw or Decrease Steroids
Description: Ability to withdraw or decrease steroids to ˂0.5 mg/kg of methylprednisolone or equivalent
Time Frame: From first dose of itacitinib until end of study treatment, up to 24 months
Population: Participants must have had one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Itacitinib
Number analyzed (Participants) | 15
Participants | 9

3. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined as the time from the first day of study drug administration (Day 1) to death on study. Patients who are alive will be censored at the date of last known date alive.
Time Frame: Every 3 months for 1 year after last dose of study treatment, up to 29 months.
Population: Participants must have had one dose of study drug and must have had 1 post-baseline disease evaluation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Itacitinib
Number analyzed (Participants) | 15
months | NA [15.5 to NA] — The median and upper limit of the 95% CI are not estimable by Kaplan-Meier method based on the data and events collected due to an insufficient number of participants with death events.

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events as a Measure of Safety and Tolerability of Itacitinib
Description: Adverse events will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE Version 5.0)
Time Frame: Safety will be assessed from the time that informed consent is signed until 30 days after the last dose of study treatment, up to 25 months.
Population: Participants must have had one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Itacitinib
Number analyzed (Participants) | 15
Participants | 15

5. Secondary Outcome: Number of Participants With Improvement in Quality of Life Per the Lee Symptom Scale
Description: Changes in symptom burden will be measured using the Lee Symptom Scale. Subscale scores and the summary score range from 0 to 100, with a higher score indicating worse symptoms.
Time Frame: Quality of life will be assessed prior during screening and end of treatment, up to 24 months of treatment. Participants showing improvement in LSS score from Screening to End of Treatment are shown here.
Population: Participants must have had one dose of study drug and must have had 1 post-baseline disease evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Itacitinib
Number analyzed (Participants) | 15
Participants | 11

6. Secondary Outcome: Number of Participants With Recurrence or Progression of cGVHD
Description: Participants will be assessed for severity of cGVHD using the Clinician-Reported Global cGVHD Activity Assessment Form and Patient-reported cGVHD Activity Assessment Form. Progression in at least one organ or site without a response in any other organ or site per NIH 2014 Consensus Development Project on Clinical Trials in cGVHD.
Time Frame: cGVHD status will be assessed at cycle 1 day 1, day 1 of every cycle and at the end of treatment, up to 24 months
Population: Participants must have had one dose of study drug and must have had 1 post-baseline disease evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Itacitinib
Number analyzed (Participants) | 15
Participants | 5

7. Secondary Outcome: Relapse Rate of Underlying Malignancy
Description: Participants will be closely monitored for any evidence of underlying disease relapse or recurrence. Formal re-staging will be done at physician discretion.
Time Frame: Relapse of underlying malignancy will be assessed on Day 1 of each cycle, at end of treatment and survival follow-up. Follow-up visits every 3 months for 1 year after last dose of study treatment, up to 29 months
Population: Participants must have had one dose of study drug and must have had 1 post-baseline disease evaluation.
Measure: Number; unit: participants
Arm/Group | Itacitinib
Number analyzed (Participants) | 15
participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time that informed consent is signed until 30 days after the last dose of study treatment, up to 25 months. All-Cause Mortality was assessed up to 29 months.
Description: Adverse events will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE Version 5.0)
Arm/Group | Itacitinib
All-Cause Mortality (participants affected / at risk) | 2/15
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Itacitinib (N=15)
Brain contusion (Injury, poisoning and procedural complications) | 1
Cellulitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Embolism (Vascular disorders) | 1
Eye contusion (Injury, poisoning and procedural complications) | 1
Pneumatosis (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract infection bacterial (Infections and infestations) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Itacitinib (N=15)
Anaemia (Blood and lymphatic system disorders) | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Balance disorder (Ear and labyrinth disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Cataract (Eye disorders) | 1
Cataract operation (Eye disorders) | 2
Conjunctival haemorrhage (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Vision blurred (Eye disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Oral dysaesthesia (Gastrointestinal disorders) | 1
Oropharyngeal pain (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 2
Fatigue (General disorders) | 4
Generalised oedema (General disorders) | 2
Localised oedema (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 1
Pyrexia (General disorders) | 4
Angioedema (Immune system disorders) | 1
Candida infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 3
Epstein-Barr virus infection reactivation (Infections and infestations) | 1
Food poisoning (Infections and infestations) | 1
Gram stain positive (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Polyomavirus viraemia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 3
Rib fracture (Injury, poisoning and procedural complications) | 1
Skin wound (Injury, poisoning and procedural complications) | 2
Wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 3
Blood cholesterol increased (Investigations) | 3
Blood creatinine increased (Investigations) | 5
Blood lactate dehydrogenase increased (Investigations) | 3
Blood lactic acid increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 3
Blood urea increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Low density lipoprotein increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Monocyte count increased (Investigations) | 1
Neutrophil count increased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Platelet count increased (Investigations) | 1
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 2
White blood cell count increased (Investigations) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypertransaminasaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypoaesthesia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Physical deconditioning (Musculoskeletal and connective tissue disorders) | 1
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 1
Orthostatic hypotension (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 3
Restless legs syndrome (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 3
Dysuria (Renal and urinary disorders) | 1
Glomerular filtration rate decreased (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 3
Erectile dysfunction (Reproductive system and breast disorders) | 1
Hypoxia (Reproductive system and breast disorders) | 3
Penile discomfort (Reproductive system and breast disorders) | 1
Vulval ulceration (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Skin laceration (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Alcohol abuse (Social circumstances) | 1
Bleeding varicose vein (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT04200365/Prot_SAP_000.pdf